CLINICAL TRIAL: NCT06494982
Title: The Influence of Augmentation of the Anterior Vaginal Wall With a Vascularized Flap on the Effectiveness of Mesh-augmented Sacrospinous Hysteropexy and Anterior Subfascial Colporrhaphy During Reconstruction of the Pelvic Floor for POP
Brief Title: The Influence of Using Vascularized Vaginal Flap on the Efficacy of Mesh-augmented Sacrospinous Hysteropexy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Shkarupa Dmitry, MD, PhD; Director, St. Petersburg State University Hospital, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vaginal flap
Record Dates: First submitted 2024-03-25; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; vaginal repair; vaginal mesh; sacrospinous fixation; vaginal flap
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacrospinous hysteropexy with the synthetic mesh, vaginal flap and anterior colporrhaphy (Active Comparator)
  Interventions: Procedure: Sacrospinous hysteropexy with the synthetic mesh, vaginal flap and anterior colporrhaphy
- Sacrospinous hysteropexy with the synthetic mesh and anterior colporrhaphy (Active Comparator)
  Interventions: Procedure: Sacrospinous hysteropexy with the synthetic mesh and anterior colporrhaphy

INTERVENTIONS:
Procedure: Sacrospinous hysteropexy with the synthetic mesh, vaginal flap and anterior colporrhaphy — Sacrospinous hysteropexy with the synthetic mesh, vaginal flap and anterior colporrhaphy
  Arms: Sacrospinous hysteropexy with the synthetic mesh, vaginal flap and anterior colporrhaphy
Procedure: Sacrospinous hysteropexy with the synthetic mesh and anterior colporrhaphy — Sacrospinous hysteropexy with the synthetic mesh and anterior colporrhaphy
  Arms: Sacrospinous hysteropexy with the synthetic mesh and anterior colporrhaphy

SUMMARY:
This is a prospective randomized controlled trial designed to compare the effectiveness and safety of two methods of pelvic floor reconstruction in patients with pelvic organ prolapse (POP): sacrospinous hysteropexy (SSHP) with synthetic mesh, vascularized anterior vaginal wall flap, anterior colporrhaphy, and sacrospinous hysteropexy with synthetic mesh. , anterior colporrhaphy, as well as the impact of surgery on quality of life.

DETAILED DESCRIPTION:
BACKGROUND POP is an epidemiologically widespread condition, occurring in 40-60% of women who have given birth. With all the variety of anatomical defects of the pelvic floor, the most common variant is prolapse of the anterior vaginal wall (cystocele).

Of the currently known surgical methods for the treatment of cystocele, anterior colporrhaphy occupies one of the most key places. However, the high recurrence rate of 7-23%, and according to some authors more than 90%, has led to the development of new techniques. In 1997, M. Cosson proposed the "Plastron" method, the essence of which is to close the defect of the pubocervical fascia by fixing a de-epithelialized flap of the anterior vaginal wall to the tendinous arch of the pelvic fascia and then performing anterior colporrhaphy over it. The method was effective in 93.5% of cases in patients with cystocele. At the same time, apical prolapse is present in many women with cystocele. Apical support is important in maintaining normal pelvic floor anatomy. Patients who undergo anterior vaginal wall repair with concomitant repair of the apical defect have a lower risk of reoperation for POP.

There are various methods for restoring apical defects while preserving the uterus. SSHP is the most studied method and was originally performed using sutures. The use of transvaginal mesh for SSHP remains controversial due to the high risk of mesh-associated complications, although many authors report the safety and high effectiveness of the SSHP method using transvaginal mesh. Despite this, the issue of cystocele recurrence after SSHP (with or without mesh) in combination with anterior colporrhaphy remains unresolved.

PREOPERATIVE ASSESSMENT All patients who meet eligibility criteria will undergo a preoperative assessment: medical history, physical and vaginal examination, assessing pelvic organ prolapse according to Pelvic Organ Prolapse Quantification System (POP-Q). All patients will complete questionnaires validated in Russia: Pelvic Floor Disability Index (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, short form (PISQ-SF), Patient Global Impression of Improvement (PGI-I).

MATERIALS AND METHODS The investigators hypothesis is that is that the use of a deepithelialized vascularized flap of the anterior vaginal wall when performing mesh-augmented sacrospinous hysteropexy and anterior subfascial colporrhaphy reduces the risks of developing relapses of POP in the anterior compartment.

The sample size was calculated taking into account the reported rate of cystocele recurrence using each technique in the literature (6.5% for sacrospinous hysteropexy using vaginal flap vs. 38.7% for mesh-augmented sacrospinous hysteropexy using subfascial colporrhaphy). With a power of 80%, a level of 0,05 and the non-inferiority margin at 15%, the sample size is 50 patients. The investigators assume a drop-out rate of 20%, thus a total of 60 participants will be included in the study.

All enrolled patients will be randomly assigned to SSHP using mesh, vaginal flap and anterior colporrhaphy or SSHP using mesh and anterior colporrhaphy treatment groups in equal ratio the day before the surgery, using computer randomization.

All data will be collected by medical staff not involved in treatment. Collected pre- and postoperative data will be anonymized using unique codes, that patients will receive immediately after randomization.

All surgical interventions will be performed by 3 qualified surgeons. Postoperative follow-up will be performed 6 and 12 months after surgery by 2 researchers, who will be blinded about the type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a woman with anterior and apical compartment pelvic organ prolapse
* The age of a subject is 45-80 years
* Leading point of prolapse is at the level of the hymen or distal to the hymen (Ba, C>=1 according to POP-Q classification)
* The subject gave written consent to participate in the study
* The subject is able to evaluate the risks of the treatment and make an independent decision on participation in the study
* The subject is able to fill up validated questionnaires and come to the control visit after the surgery

Exclusion Criteria:

* The subject has an active urinary tract infection or skin infection in the region of surgery or acute infectious disease
* The subject had prior hysterectomy
* The subject has previously diagnosed or currently active cancer
* The subject has chronic pelvic pain
* The subject has cervical elongation
* The subject has gynecological diseases (recurrent uterine bleeding, endometrial hyperplasia, the presence of atypical cells in cervical smears, adenomyosis, multiple uterine myoma)
* The subject is planning pregnancy
* The subject is unable to visit postoperative check-ups
* Refusal from participation.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective cure rate | 12 months (1 year)
  The patient is considered cured if there is no prolapse beyond the hymen and the cervix is above -1 cm according to POP-Q (0-1 stage)

SECONDARY OUTCOMES:
Satisfaction with the surgery | Measured postoperatively at intervals of 6, 12 months postoperatively, up to 100 weeks
  Measured through the Patient Global Impression of Improvement questionnaire (PGI-I), validated in Russia. The patient marks the number that best describes her post-operative condition, compared with how it was before surgery. The score ranges from 1 (very much better) to 7 (very much worse).
The impact of treatment on sexual function | Measured postoperatively at intervals of 6, 12 months postoperatively, Measured postoperatively at intervals of 6, 12 months postoperatively, up to 100 weeks
  Measured through the scoring of Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) validated in Russia. The scale evaluates sexual function in patients with urinary incontinence and/or POP. The responses are graded on a five-point Likert scale ranging from 0 (always) to 4 (never). Items 1 - 4 are reversely scored and a total of 48 is the maximum score. The higher scores indicate better sexual function.
The impact of treatment on the quality of life | Measured postoperatively at intervals of 6, 12 months postoperatively, Measured postoperatively at intervals of 6, 12 months postoperatively, up to 100 weeks
  Measured through the Pelvic Floor Disability Index (PFDI-20), validated in Russia. The item includes 20 questions. The score ranges from 0 to 300. The higher the score, the worse the outcome.
Observed complications | Measured postoperatively at intervals of 6, 12 months postoperatively, Measured postoperatively at intervals of 6, 12 months postoperatively, up to 100 weeks
  Presence of any adverse effects such as: bleeding requiring blood transfusion, haematoma, organ perforation, nerve injury, vaginal scarring and shortening, wound infection, urinary tract infection, pelvic pain, mesh extrusion in the vagina, mesh erosion into the urinary tract, dyspareunia de novo, de novo urgency, atonic bladder, de novo stress urinary incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Shkarupa, MD, PhD, Study Chair — Saint Petersburg State University, Russia
Locations (1):
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No